CLINICAL TRIAL: NCT03016026
Title: Effect of Enhanced Recovery After Surgery (ERAS) on Laparoscopy-assisted Distal Subtotal Gastrectomy: A Single Arm Trial
Brief Title: Enhanced Recovery After Surgery (ERAS) on Laparoscopy-assisted Distal Gastrectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Guoxin Li, M.D.,Ph.D., Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERAS-LAG-01
Record Dates: First submitted 2016-11-24; First posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Stomach Neoplasms
Keywords: ERAS,Laparoscopy,Distal Gastrectomy,Safety,Effectiveness
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ERAS (Experimental): Preoperative education,breathing training and atomizing during the time of preoperative preparation.Shorten fasting time and carbohydrate load.The intravenous fluid therapy is restricted.Drainage and nasogastric tube are not placed (except the concerns of surgical safety).All patients undergo laparoscopic distal gastrectomy.An optimal management of acute postoperative pain is multimodal analgesia consists of surgical site infiltration, a nonsteroidal anti-inflammatory drug for postoperative three days (POD) and epidural analgesia.Early oral take and move.
  Interventions: Procedure: ERAS

INTERVENTIONS:
Procedure: ERAS — Undergo an ERAS program

SUMMARY:
This study evaluates the safety and effectiveness of enhanced recovery after surgery(ERAS) on laparoscopic distal gastrectomy for gastric cancer.All of participants received an ERAS program.

DETAILED DESCRIPTION:
Preoperative education about ERAS program is administered in the ward after admission by a specific team. Breathing training and atomizing during the time of preoperative preparation is performed during hospitalization (5-7 days). Patients are allowed to eat a normal diet and intake of 1000 ml 10% carbohydrate drink 10 hours before surgery and oral 500ml 10% carbohydrate drink 2 hours before the induction of anesthesia. Mechanical bowel preparation is not recommended as routine procedure.

The intravenous fluid therapy is restricted. Urinary catheters are routinely placed after anesthesia. In principle, drainage and nasogastric tube are not placed (except the concerns of surgical safety). Surgical site infiltration is implemented.All patients undergo laparoscopic distal gastrectomy.

Urinary catheters are routinely removed within 24 hours after operation. An optimal management of acute postoperative pain is multimodal analgesia consists of surgical site infiltration, a nonsteroidal anti-inflammatory drug for postoperative three days (POD) and epidural analgesia. Adjunctive analgesia with acetaminophen is used after the resumption of oral intake until adequate pain relief. Patients were encouraged to move from POD 1. The patients are encouraged to a full fluid diet on POD 2. Adhere to the premise of eating little and often daily increase, then to semi-fluids to soft diet. A normal diet is often started on POD 4. Abdominal drains are routinely removed within 72 hours after operation.

ELIGIBILITY:
Inclusion Criteria:

* Age from over 18 to under 75 years
* Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
* cT1-4a, N0-3, M0 at preoperative evaluation according to the AJCC Cancer Staging Manual Seventh Edition
* Expected curative resection through distal subtotal gastrectomy with D2 lymphadenectomy
* no severe organ dysfunction
* Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale
* ASA (American Society of Anesthesiology) score class I or II
* Written informed consent

Exclusion Criteria:

* Women during pregnancy or breast-feeding
* Severe mental disorder
* History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
* History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
* Enlarged or bulky regional lymph node diameter over 3cm by preoperative imaging
* History of other malignant disease within past five years
* History of previous neoadjuvant chemotherapy or radiotherapy
* History of unstable angina or myocardial infarction within past six months
* History of cerebrovascular accident within past six months
* History of continuous systematic administration of corticosteroids within one month
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* FEV1<50% of predicted values

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative hospital stays | 1 month
  Days from surgery to discharge
Rehabilitative rate | 4 days
  Postoperative 4 days

SECONDARY OUTCOMES:
Medical cost | 1 month
  From surgery to discharge
Postoperative pain score | 4 days
  Postoperative 4 days
Postoperative recovery index | 1 month
Postoperative inflammatory immune response | 4 days
  Postoperative 4 days
Morbidity rates | 30 days
Mortality rates | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Guoxin Li, MD.,Ph.D, Principal Investigator — Southern Medical University, Guangzhou,China; Kexuan Liu, MD.,Ph.D, Principal Investigator — Southern Medical University, Guangzhou,China; Hao Liu, MD.,Ph.D, Study Director — Southern Medical University, Guangzhou,China; Li Zhen, MD.,Ph.D, Study Director — Southern Medical University, Guangzhou,China; Xiaomin Hou, MD.,Ph.D, Study Director — Southern Medical University, Guangzhou,China; Jiang Yu, MD.,Ph.D, Study Director — Southern Medical University, Guangzhou,China; Yu Zhu, MD., Study Director — MD.,Ph.D
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liang Y, Liu H, Nurse LZ, Zhu Y, Zhao M, Hu Y, Yu J, Li C, Liu K, Li G. Enhanced recovery after surgery for laparoscopic gastrectomy in gastric cancer: A prospective study. Medicine (Baltimore). 2021 Feb 19;100(7):e24267. doi: 10.1097/MD.0000000000024267. PMID 33607765